CLINICAL TRIAL: NCT02155829
Title: Riluzole for PTSD: Efficacy of a Glutamatergic Modulator as Augmentation Treatment for Posttraumatic Stress Disorder
Brief Title: Safety Study of Riluzole to Treat Post-traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, David M. Benedek, Principal Investigator, Uniformed Services University of the Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 380797
Record Dates: First submitted 2013-11-15; First posted 2014-06-04 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: PTSD
Keywords: PTSD; TBI; Riluzole; Rilutek; augmentation; supplement; double blinded; clinical trial; placebo; RCT; Randomized Control Trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Riluzole; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Riluzole (Experimental): Weeks 1 and 2: Riluzole 50 mg tablet by mouth every 12 hours (100 mg/day) for 2-weeks
  Weeks 3 to 8 (optional dose increase): 2 Riluzole 50 mg tablets by mouth every 12 hours (200 mg/day) for 6-weeks
  Interventions: Drug: Riluzole
- Placebo (Placebo Comparator): Weeks 1 and 2: Placebo 50 mg tablet by mouth every 12 hours (100 mg/day) for 2-weeks
  Weeks 3 to 8 (optional dose increase): 2 Placebo 50 mg tablets by mouth every 12 hours (200 mg/day) for 6-weeks
  Interventions: Drug: Placebo (for Riluzole)

INTERVENTIONS:
Drug: Riluzole
  Other Names: Rilutek
  Arms: Riluzole
Drug: Placebo (for Riluzole)
  Other Names: Inert tablet manufactured to be indistinguishable from a Riluzole 50 mg tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Riluzole is effective in the augmentation treatment of post-traumatic stress disorder (PTSD) that is experienced by Active Duty military service members and Operation Enduring Freedom (OEF), Operation Iraqi Freedom (OIF), and Operation New Dawn (OND) veterans who have not had symptom reduction after one or more kinds of medications or therapies.

DETAILED DESCRIPTION:
Riluzole is a glutamatergic modulator that inhibits glutamate release and enhances AMPA trafficking and clearance of excessive synaptic glutamate resulting in neuroprotective properties. Riluzole is FDA-approved for the treatment of amyotrophic lateral sclerosis (ALS) and has been found to have antidepressant and anxiolytic properties in animals and in humans (Zarate et al., 2004). Posttraumatic stress disorder (PTSD) is a chronic and seriously debilitating anxiety disorder that develops following exposure to severe trauma, such as combat exposure. Structural magnetic resonance imaging has been used to measure the volume of crucial structures implicated in the pathophysiology of PTSD, with several morphometric studies confirming smaller hippocampal volume in PTSD patients. Current pharmacological treatment for PTSD, and particularly combat-related PTSD, is suboptimal. Drugs that alter neuronal survival pathways through reduction of glutamate activity may play a role in reversing the loss of neuronal integrity and possible focal atrophy in regions of the brain implicated in the pathophysiology of PTSD, potentially improving the symptoms of PTSD, as well as TBI. This study will evaluate the efficacy of acute riluzole treatment in active duty and Operation Iraqi Freedom (OIF), Operation Enduring Freedom (OEF), and Operation New Dawn (OND) veterans with PTSD, with or without mild TBI (mTBI), who are sub-optimally responsive to other medication treatments. A total of 158 active duty and OIF, OEF and OND veterans, aged 18 to 65 will be enrolled from WRNMMC and the Syracuse VA Medical Center to participate in this 8-week randomized, double- blind, placebo-controlled, parallel study. Patients who are suboptimal responders to their current psychotropic drugs will continue these at stable dosage for at least 2 weeks prior to randomization during the screening period. We hypothesize that those subjects with PTSD, with or without mTBI, who are only partially responsive to initial therapy and are subsequently randomized to augmentation therapy with Riluzole (100-200mg/day) will have a superior response rate compared to those subjects randomized to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Active-duty service member or an Operation Iraqi Freedom (OIF), Operation Enduring Freedom (OEF), or Operation New Dawn (OND) veteran.
* Clinical diagnosis of PTSD and have not achieved remission with an adequate trial of medication treatment (8 weeks) as indicated by self-report at referral and confirmed by baseline CAPS score of greater than or = to 40 after informed consent is obtained.

Exclusion Criteria:

1. Female subjects of childbearing capacity who test positively for ß-HCG, or are either self-reporting as pregnant, planning to become pregnant, or nursing.
2. Presence of psychotic features.
3. Unable to provide informed consent or comply with study procedures.
4. Previous treatment with riluzole.
5. Serious, unstable illnesses including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, hematologic disease, or HIV. This includes individuals with a history of COPD by diagnosis as well as persons taking inhalers for Asthma or Reactive Airway Disease.
6. Clinically significant abnormal levels (3x ULN or greater) of serum transaminases (ALT/SGPT; AST/SGOT), current or past blood dyscrasia.
7. Subjects with uncorrected hypothyroidism or hyperthyroidism.
8. DSM-IV alcohol or substance abuse or dependence within 90 days of the screening visit.
9. Treatment with a reversible MAOI, guanethidine, or guanadrel within 1 week, or any change in fluoxetine dosing within 8 weeks prior to visit 2. Use of antidepressant and sedative/hypnotic drugs at stable dose is permitted.
10. Documented history of hypersensitivity or intolerance to riluzole.
11. Subjects with a current or past history of other axis I disorders including schizophrenia, schizoaffective disorder, bipolar disorder or dementia. However, those with a co-morbid history of other Axis I disorder like major depression, dysthymia or other anxiety disorders will be included; the justification for this is that approximately 70% of subjects with PTSD have co-morbid depression and or alcohol abuse, and restricting the sample to PTSD patients without depression will not accurately reflect the scope of this disorder.
12. Patients who are currently at high risk for homicide or suicide, as indicated by an affirmative answer to the question: "In the last three months, have you attempted to kill yourself, made specific plans to kill yourself, or had the intention to kill yourself?"
13. Current or planned litigation regarding the traumatic event.
14. Patients who recently started trauma focused cognitive behavioral psychotherapy (Patient's underlying educational or supportive individual or group therapy will be included).
15. Patient's actively enrolled in an evidence based psychotherapy treatment (e.g., Cognitive Processing Therapy or Prolonged Exposure Therapy) will be excluded until that therapy has concluded, but may be re-approached at that time if patient self-report or clinician referral suggests persistent PTSD symptoms upon conclusion of that treatment.
16. Subjects with an artificial cardiac pacemaker or metallic implants within their body will be enrolled at WRNMMC for the placebo-control clinical trial portion of the study only. These individuals, due to their pre-existing medical condition, are medically ineligible to participate in the 1H MRS imaging portion of the study. Further, the Magnetic Resonance (MRI) Screening Form is use at WRNMMC will be used for participant screening prior to any imaging procedures.
17. Use of benzodiazepines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-07; Primary Completion 2017-10-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Benedek, MD, Principal Investigator — USUHS, WRNMMC
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Syracuse VA Medical Center, Center for Integrated Healthcare (116C), Syracuse, New York

REFERENCES:
- [Derived] Spangler PT, West JC, Dempsey CL, Possemato K, Bartolanzo D, Aliaga P, Zarate C, Vythilingam M, Benedek DM. Randomized Controlled Trial of Riluzole Augmentation for Posttraumatic Stress Disorder: Efficacy of a Glutamatergic Modulator for Antidepressant-Resistant Symptoms. J Clin Psychiatry. 2020 Oct 27;81(6):20m13233. doi: 10.4088/JCP.20m13233. PMID 33113596
- See also: Study conducted by the Center for the Study of Traumatic Stress — http://www.cstsonline.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from WRNMMC = Walter Reed National Military Medical Center ; SVAMC = Syracuse Veterans Administration Medical Center
Period: Overall Study
Arm/Group | Riluzole | Placebo
Started | 37 | 38
Completed | 31 | 35
Not Completed | 6 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: One participant failed to meet minimum Clinician-Administered PTSD Scale IV (CAPS-IV) score for inclusion at phase 2 baseline and was excluded from intent-to treat (ITT) analyses.
Groups:
- Riluzole: Weeks 1 and 2: Riluzole 50 mg tablet by mouth every 12 hours (100 mg/day) for 2-weeks
  Weeks 3 to 8 (optional dose increase): 2 Riluzole 50 mg tablets by mouth every 12 hours (200 mg/day) for 6-weeks
  Riluzole
- Placebo: Weeks 1 and 2: Placebo 50 mg tablet by mouth every 12 hours (100 mg/day) for 2-weeks
  Weeks 3 to 8 (optional dose increase): 2 Placebo 50 mg tablets by mouth every 12 hours (200 mg/day) for 6-weeks
  Placebo (for Riluzole)
- Total: Total of all reporting groups
Arm/Group | Riluzole | Placebo | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (8.9) | 38.1 (8.2) | 37.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 31 | 32 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 3 | 12
  Not Hispanic or Latino | 23 | 33 | 56
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 2 | 6 | 8
  White | 26 | 25 | 51
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 4 | 3 | 7
Clinician Administered PTSD Scale - IV [Mean (Standard Deviation); unit: units on a scale] — A summed score of 17 items.
  Minimum Score: 0 (no symtpoms)
  Maximum Score: 136 (very severe symptoms)
  Subscales:
  Subscale B (re-experiencing): items 1-5, a score of 0-40. Subscale C (avoidance): items 6-12, a score of 0-56. Subscale D (hyperarousal): items 13-17, a score of 0-40.
  units on a scale | 70.6 (19.8) | 62.4 (16.9) | 66.4 (18.7)

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale (CAPS) Score
Description: CAPS is a 30-item structured interview that can be used to make current (past month) diagnoses of PTSD, make lifetime diagnoses of PTSD, and assess PTSD symptoms over the past week.
  A summed score of 17 items:
  Minimum Score: 0 (no symptoms)
  Maximum Score: 136 (very severe symptoms)
  Subscales:
  Subscale B (re-experiencing): items 1-5, a score of 0-40. Subscale C (avoidance): items 6-12, a score of 0-56. Subscale D (hyperarousal): items 13-17, a score of 0-40.
  CAPS scores were measured at baseline, mid-treatment, and post-treatment. For outcome analyses, differences between pre-treatment and post-treatment scores were used.
Time Frame: Week 1 and 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 36 | 38
score on a scale | -21.1 (18.9) | -16.7 (17.2)
Statistical Analysis 1: Comparison: Riluzole vs Placebo; Test type: Superiority; p = 0.442, ANCOVA; ANCOVA covariate included site

2. Secondary Outcome: PTSD Check List Specific (PCL-S)
Description: A 17-item self-report measure used to assess PTSD symptoms related to a specific traumatic event.
  Scoring: A sum of all 17 items. Minimum: 17 (no symptoms) Maximum: 85 (very severe symptoms)
  PCL-S scores were measured at every study visit. For outcome analyses, differences between pre-treatment and post-treatment scores were used.
Time Frame: Week 1 and 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 36 | 38
score on a scale | -15.4 (13.5) | -14.5 (11.4)
Statistical Analysis 1: Comparison: Riluzole vs Placebo; Test type: Superiority; p = 0.994, ANCOVA; ANCOVA covariate included site

3. Secondary Outcome: Montgomery-Åsberg Depression Rating Scale (MADRS) Score
Description: A ten-item diagnostic questionnaire to measure the severity of depressive episodes.
  Scoring: A sum of all 10 items. Minimum: 0 (no symptoms) Maximum: 60 (very severe symptoms)
  MADRS scores were measured at every study visit. For outcome analyses, differences between pre-treatment and post-treatment scores were used.
Time Frame: Week 1 and 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 36 | 38
score on a scale | -7.9 (7.6) | -8.2 (9.6)
Statistical Analysis 1: Comparison: Riluzole vs Placebo; Test type: Superiority; p = 0.684, ANCOVA; ANCOVA covariate included site

4. Secondary Outcome: Hamilton Anxiety Rating Scale (HAM-A)
Description: A 14-item clinician-administered assessment measuring anxiety symptoms.
  Scoring: A sum of all 14 items. Minimum: 0 (no symptoms) Maximum: 56 (very severe symptoms)
  HAM-A scores were measured at baseline, mid-treatment, and post-treatment. For outcome analyses, differences between pre-treatment and post-treatment scores were used.
Time Frame: Week 1 and 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 36 | 38
score on a scale | -7.8 (7.4) | -6.7 (6.9)
Statistical Analysis 1: Comparison: Riluzole vs Placebo; Test type: Superiority; p = 0.913, ANCOVA; ANCOVA covariate included site

5. Secondary Outcome: Sheehan Disability Scale (SDS) Score
Description: A 3-item self-report measure to assess functional impairment in work/school, social, and family life.
  Scoring: A sum of all 3 items. Minimum: 0 (no symptoms) Maximum: 30 (very severe symptoms)
  SDS scores were measured at baseline, mid-treatment, and post-treatment. For outcome analyses, differences between pre-treatment and post-treatment scores were used.
Time Frame: Week 1 and 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 36 | 38
score on a scale | -6.3 (6.8) | -5.7 (5.9)
Statistical Analysis 1: Comparison: Riluzole vs Placebo; Test type: Superiority; p = 0.746, ANCOVA; ANCOVA covariate included site

6. Secondary Outcome: Clinician Administered PTSD Subscale D (CAPS-D)
Description: Subscale D (items 13-17 on the CAPS-IV) measures Hyperarousal symptoms of PTSD
  Scoring: A sum of items 13-17. Minimum: 0 (no symptoms) Maximum: 40 (very severe symptoms)
  CAPS-D scores were measured at baseline, mid-treatment, and post-treatment. For outcome analyses, differences between pre-treatment and post-treatment scores were used.
Time Frame: Week 1 and 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 36 | 38
score on a scale | -6.8 (8.2) | -3.7 (7.3)
Statistical Analysis 1: Comparison: Riluzole vs Placebo; Test type: Superiority; p = 0.057, ANCOVA; ANCOVA covariate included site

7. Secondary Outcome: PTSD Checklist - D (PCL-D)
Description: The subscale D (items 13-17 on the PCL) measures hyperarousal symptoms of PTSD. Scoring: A sum of items 13 to 17. Minimum: 5 (no symptoms) Maximum: 25 (very severe symptoms)
  PCL-D scores were measured at baseline, mid-treatment, and post-treatment. For outcome analyses, differences between pre-treatment and post-treatment scores were used.
Time Frame: Week 1 and week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 36 | 38
score on a scale | -5.9 (5.6) | -3.4 (4.9)
Statistical Analysis 1: Comparison: Riluzole vs Placebo; Test type: Superiority; p = 0.0496, ANCOVA; ANCOVA covariate included site

8. Other Pre Specified Outcome: NAA/Cr Ratio
Description: The N-acetyl aspartate to creatine ratio (NAA/Cr) in the hippocampus and anterior cingulate, measured using magnetic resonance spectroscopy (1H MRS), will be evaluated for change after 8-week treatment with riluzole.
Time Frame: Measured at study start (Week 0) for baseline and measured at study completion (Week 8)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Riluzole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 2/37 | 0/38
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riluzole (N=37) | Placebo (N=38)
Gastrointestinal Symptoms (Gastrointestinal disorders) | 2 (2) | 0 (0) — AE resulting in drug dose reduction or emergency medical care: n = 2 Both participants were on active drug, and both reported gastrointestinal symptoms.
LFT Elevation (Hepatobiliary disorders) | 2 (2) | 0 (0) — elevation of AST/ALT greater than 3X normal
Clinical deterioration (Psychiatric disorders) | 1 (1) | 0 (0) — worsening of symptoms resulting in hospitalization

LIMITATIONS AND CAVEATS:
Result limited to combat-related PTSD in military and veterans of recent conflict.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT02155829/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT02155829/ICF_001.pdf